CLINICAL TRIAL: NCT00131144
Title: A Randomized, Controlled Study on the Efficacy and Safety of Octreotide Acetate in Microspheres in the Therapy of Patients With Moderately Severe or Severe Non-proliferate Diabetic Retinopathy (NPDR) or Low Risk Proliferative Diabetic Retinopathy (PDR)
Brief Title: Octreotide Acetate in Microspheres in Patients With Diabetic Retinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSMS995 0802
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy,Octreotide Acetate in Microspheres
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Octreotide; Microspheres

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Octreotide Acetate in Microspheres 20 mg (Experimental): 20 mg will be administered im once every 4 weeks
  Interventions: Drug: Octreotide Acetate in Microspheres 20 mg
- Octreotide Acetate in Microspheres 30 mg (Experimental): 30 mg will be administered im once every 4 weeks
  Interventions: Drug: Octreotide Acetate in Microspheres
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide Acetate in Microspheres 20 mg
  Arms: Octreotide Acetate in Microspheres 20 mg
Drug: Octreotide Acetate in Microspheres
  Arms: Octreotide Acetate in Microspheres 30 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The most common ocular disease in patients with diabetes, diabetic retinopathy, is present in approximately 40% of diabetic patients; about 8% of diabetic patients have vision threatening diabetic retinopathy. Although intensive control of blood glucose has been shown to reduce the development and progression of diabetic retinopathy, intensive control of glucose is usually not achieved in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with type 1 and type 2 diabetes mellitus
* Moderately severe or severe NPDR or mild PDR in at least one eye:

  * with an Early Treatment Diabetic Retinopathy Study (ETDRS) visual score of > 35 letters; and
  * not previously treated with scatter photocoagulation.
* HbA1c < 13% at study entry

Exclusion Criteria:

* Condition which could interfere with the assessment of retinopathy progression
* History of symptomatic gallstones without cholecystectomy
* Brittle diabetes or history of severe hypoglycemia unawareness
* Previous treatment with a somatostatin analogue

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 1999-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
time to progression of diabetic retinopathy | throughout study

SECONDARY OUTCOMES:
time to development or progression of macular edema, and | Baseline through end of study
time to moderate vision loss | Baseline through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — East Hanover
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Pivonello R, Muscogiuri G, Holder G, Paul M, Sarp S, Lesogor A, Jordaan P, Eisinger J, Colao A. Long-term safety of long-acting octreotide in patients with diabetic retinopathy: results of pooled data from 2 randomized, double-blind, placebo-controlled phase 3 studies. Endocrine. 2018 Apr;60(1):65-72. doi: 10.1007/s12020-017-1448-5. Epub 2017 Nov 7. PMID 29116540